CLINICAL TRIAL: NCT07161986
Title: Mapping Relapse Risk and Evaluating an Integrated Approach for Preventing Relapse in Polydrug Users: A Randomized Control Trial
Brief Title: Mapping And Preventing Relapse Risk in Polydrug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychology, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H24149; 2021ZD0202104 (Other Grant/Funding Number: Center for Excellence in Brain Science and Intelligence Technology)
Record Dates: First submitted 2025-08-24; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Drug Addiction; Polysubstance Addiction
Keywords: Illicit Drug use; Relpase Prevention; Mindfullness intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study consist of two groups, one is taking mindfullness intervention and other is Treatment as Usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfullness Based Intervention (Active Comparator): Mindfullness based intervention arm is taking intervention which is based on Mindfullness based sobriety manaual for Relpase prevention and craving as primary outcome
  Interventions: Behavioral: Mindfullness based Sobriety (MBS)
- Treatment As Usual (No Intervention): Treatment as usual group would take tradational treatment at rehablitataion center not particular intervention

INTERVENTIONS:
Behavioral: Mindfullness based Sobriety (MBS) — MBS is combination of Mindfullness , Relapse prevention, motivational interviewing , acceptance and commitment therapy. It helps in dealing underlying depression and anxiety issues among Polysubstance use. it Cover most of underlying problem faced by person with addiction.
  Arms: Mindfullness Based Intervention

SUMMARY:
This Interventional two-arm comparative study will evaluate whether a mindfulness-based strategy (MBS) improves outcomes for adults with substance use disorders (polydrug users) compared with treatment-as-usual (TAU). The primary question is whether MBS lowers cravings and reduces relapse risk relative to TAU; secondary aims include improvements in emotion regulation, coping, depressive/anxiety symptoms, mindfulness, and motivation to change. The design includes two arms (MBS vs TAU) with baseline and post-intervention assessments; adherence within the MBS arm will also be examined (e.g., high- vs low-adherence) to test whether greater adherence yields better primary and secondary outcomes than TAU. Primary outcomes are craving and relapse risk; secondary outcomes are emotion regulation, coping, depressive and anxiety symptoms, mindfulness, and motivation to change. Hypotheses predict that MBS will reduce cravings and depressive/anxiety symptoms and improve mindfulness and emotion regulation as compared to TAU; that psychological network structure will differ by relapse-risk level and by adherence subgroup; and that motivation to change will mediate MBS effects.

DETAILED DESCRIPTION:
This prospective observational, two-arm comparative study is to evaluate whether a mindfulness-based strategy (MBS) improves clinical and psychosocial outcomes and reduces relapse risk among adults with substance use disorders (polydrug users). The main question is whether long-term participation in MBS lowers cravings and reduces relapse risk compared with treatment-as-usual (TAU). The design includes two arms-an MBS arm (participants receiving the mindfulness-based strategy as part of care) and a TAU arm (participants receiving treatment as usual)-with adherence to MBS also analyzed (e.g., high- vs low-adherence subgroups). Participants will be adults with SUDs/polydrug use; the target sample size is 130 Participants with MBS (n=60) and TAU (n=70). Baseline and post-intervention assessments were conducted, using measures culturally adapted to Urdu. The objectives are to test whether MBS reduces substance cravings and relapse risk relative to TAU; assess improvements in emotion regulation, coping, mindfulness, depression, anxiety, and motivation to change; examine how adherence to MBS relates to outcomes; and use network analysis to characterize connections among psychological variables and compare structures by relapse risk, adherence level. The hypotheses are: H1 (Primary/Secondary): MBS will reduce cravings and Relapse Risk (primary) and depressive/anxiety symptoms, improve mindfulness, motivation to Change and emotion regulation (secondary). H2 (Primary/Secondary): Higher MBS adherence will yield better primary (Reduce craving, relapse risk) and secondary outcomes than TAU. H3: Network density/connectivity among psychological variables will differ by relapse-risk level within MBS. H4: Post-test network structures will differ between high- vs low-adherence MBS participants. H5: The Study 2 network will show weaker links between relapse factors and symptoms than Study 1, reflecting MBS impact. H6: MBS will improve coping skills, emotion regulation, and mindfulness. H7: Motivation to change will mediate the relationship between MBS participation and outcomes. Primary outcomes are craving and relapse risk (Relapse Risk Scale; subscales: compulsivity to use, abstinence-violation effect, anxiety problems, low self-efficacy). Secondary outcomes include emotion regulation (CERQ: self-blame, acceptance, rumination, positive refocusing, planning, positive reappraisal, putting into perspective, catastrophizing, other-blame), mindfulness (MAAS; note that higher scores indicate lower mindfulness ), depression, anxiety, and stress (DASS-21), coping (Brief COPE Urdu: emotion-focused, avoidance-focused, problem-focused), and motivation to change (RCQ: precontemplation, contemplation, action). Analytically, group comparisons will contrast MBS versus TAU on primary and secondary outcomes with stratification by MBS adherence; network analysis will compare network density and structure across relapse-risk strata, adherence subgroups, and between Study 2 and Study 1; and mediation models will test whether motivation to change mediates MBS effects on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals resided in Drug rehabilitations center with polysubstance use diagnosed particularly with illicit drug use.
* Age would be from 18 to 85 years
* Must include Patients after detox and withdrawal symptoms.

Exclusion Criteria:

• Individuals with any form of physical or intellectual disability will not be eligible to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Relpase Risk | From Enrollment to end of treatment at 6 weeks and then 2 week followup
  Relapse Risk Relapse risk will be measured using the Relapse Risk Scale, consisting of four subscales: compulsivity to use, abstinence violation effect, anxiety problems, and low self-efficacy. Scores classify risk as: High (>170), Moderate (98-170), or Low (<98).
Craving | From Enrollment to end of treatment at 6 weeks and then 2 week followup
  Craving Craving will be measured using a rating scale from 1 (minimum) to 10 (maximum), with higher scores indicating greater craving intensity.

SECONDARY OUTCOMES:
Emotional Regulation Skills | From Enrollment to the end of treatment at 6 week and 2 week followup
  Measured using the Cognitive Emotion Regulation Questionnaire (Shahzad et al., 2022). Subscales include self-blame, acceptance, rumination, positive refocusing, planning, reappraisal, perspective, catastrophizing, and other-blame. Each subscale ranges from 4-20; total score ranges from 36-180. Higher scores indicate greater use of that strategy.
mental Health Conditions | From Enrollment to the end of treatment at 6 week and 2 week followup
  mental health condition such as Depression, Anxiety, and Stress will be measured using the DASS-21 (Aslam & Kamal, 2017). Scores range: Depression (0-4), Anxiety (0-3), Stress (0-7). Higher scores reflect greater symptom severity
Mindfulness (MAAS) | From Enrollment to the end of treatment at 6 week and 2 week followup
  Mindfulness Attention Awareness Scale (Bakhteyar et al., 2021). Higher scores (closer to 6) indicate higher levels of mindfulness.
Motivation to Change (RCQ) | From Enrollment to the end of treatment at 6 week and 2 week followup
  Measured via Readiness to Change Questionnaire (Mubashir et al., 2025). Subscales: Precontemplation, Contemplation, Action. Subscale scores are calculated by summing the respective item scores and high scores indicate strong identification with that specific stage of change.

OTHER OUTCOMES:
Coping Skills | From Enrollment to end of treatment at 6 weeks and then 2 week followup
  while Brief Coping Orientation of problems experienced Urdu Scale for coping skills will be used (Nisa & Siddiqui, 2020). Subscales: (emotion-focused coping, avoidance-focused coping, and problem-focused coping).Higher Scoring on subscale indicate a greater use of that specific coping. 0 to 8 with higher scores demonstrate more prominant utilization and low scores demonstrate less utilization of each coping strategies

CONTACTS AND LOCATIONS:
Overall Officials: Li Yonghui Professor, Institute Of Psychology,Chinese Acedmy of Sciences, Study Chair — Institute Of Psychology,Chinese Acedmy of Sciences; Romana Younas PhD fellow, Mphil ClPsy, Principal Investigator — Institute of Psychology,Chinese Acedmy Of Sciences; Salman Shahzad Professor, Study Director — Institute of Clinical Psychology,Universitry of Karachi,Pakistan
Locations (1):
- Save Life Foundation, Abbottābād, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
As clients are not agreed to share thier data with other party , beacsue data is confidential and bound to follow ethical consideration and regulations.

REFERENCES:
- [Background] Priddy SE, Howard MO, Hanley AW, Riquino MR, Friberg-Felsted K, Garland EL. Mindfulness meditation in the treatment of substance use disorders and preventing future relapse: neurocognitive mechanisms and clinical implications. Subst Abuse Rehabil. 2018 Nov 16;9:103-114. doi: 10.2147/SAR.S145201. eCollection 2018. PMID 30532612